CLINICAL TRIAL: NCT02734212
Title: Reducing Internalized Stigma Among Veterans With PTSD: A Pilot Trial
Brief Title: Ending Self Stigma for PTSD
Acronym: ESS-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1432-P; 1I21RX001432-01 (NIH)
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Stigmatization
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stereotyping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors were blind with regards to participants condition
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ending Self-Stigma for PTSD (Experimental): Ending Self Stigma for PTSD (ESS-P) is a 9-session small-group (6-8 persons) course designed to help individuals with PTSD develop skills to effectively cope with stigma and minimize the internalization of stigmatizing beliefs and stereotypes. Sessions combine in-class lecture, discussion of relevance to group members' personal experiences, review and practice of strategies and skills, and group sharing, support, and problem-solving. Each session is designed to focus on a specific strategy for addressing self-stigma.
  Interventions: Behavioral: Ending Self Stigma for PTSD
- Enhanced Treatment as Usual (Other): The comparison condition will consist of providing a pamphlet that discusses societal stigma and internalized stigma, and provides resources to help combat the effects of both. Participants will be given the informational pamphlet and study staff will discuss its content with the participant.
  Interventions: Other: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: Ending Self Stigma for PTSD — Ending Self Stigma for PTSD (ESS-P) is a 9-session small-group (6-8 persons) course designed to help individuals with PTSD develop skills to effectively cope with stigma and minimize the internalization of stigmatizing beliefs and stereotypes. Sessions combine in-class lecture, discussion of relevance to group members' personal experiences, review and practice of strategies and skills, and group sharing, support, and problem-solving. Each session is designed to focus on a specific strategy for addressing self-stigma.
  Other Names: ESS-P
  Arms: Ending Self-Stigma for PTSD
Other: Enhanced Treatment as Usual — The comparison condition will consist of providing a pamphlet that discusses societal stigma and internalized stigma, and provides resources to help combat the effects of both. Participants will be given the informational pamphlet and study staff will discuss its content with the participant.
  Other Names: ETAU
  Arms: Enhanced Treatment as Usual

SUMMARY:
Veterans with PTSD report that stigma and fear of stigma have a chilling effect on their participation in mental health treatment. Despite the widely-documented effects of stigma on the recovery of individuals with mental illnesses and research demonstrating harmful consequences of internalized stigma, including decreased hope, self-esteem, personal motivation, and persistence regarding illness management, no interventions are currently available to assist Veterans with PTSD in combating the impact of internalized stigma. The goal of this research is to develop and pilot-test an intervention to provide Veterans with PTSD the skills to cope effectively with stigma and to mitigate the internalization of stigmatizing beliefs and stereotypes. To accomplish this purpose, Ending Self Stigma (ESS), an intervention composed of evidence-based methods for combating internalized stigma for serious mental illness, will be modified and tested to address issues particular to PTSD.

DETAILED DESCRIPTION:
Stigma and fear of stigma are widespread among Veterans with PTSD and both have pernicious effects on Veterans' well-being and participation in mental health treatment. Internalized stigma is a harmful consequence of societal stigma, and has been associated with decreased hope, self-esteem, personal motivation, morale, self-regard, and persistence regarding illness management among individuals with a range of mental illnesses. Internalized stigma also has negative impacts on the recovery and well-being of Veterans with PTSD specifically, but no evidence-based interventions are currently available to assist Veterans with PTSD in combatting the impact of internalized stigma. Therefore, the purpose of this proposal is to develop and pilot-test an intervention to provide Veterans with PTSD the skills to cope effectively with stigma and to mitigate the internalization of stigmatizing beliefs and stereotypes. To that end, the investigators will modify Ending Self Stigma (ESS), an intervention composed of evidence-based strategies for combating internalized stigma for mental illness developed by the investigators' team, to specifically serve the needs of Veterans with PTSD.

This proposed project is composed of two phases. In Phase I, the investigators will produce an intervention and accompanying manual for the PTSD version of ESS (ESS-P), based upon the strategies and structure of the existing ESS intervention. To this end, the investigators will interview Veterans with a PTSD diagnosis to learn more about their experience with societal and internalized stigma associated with PTSD, plus other considerations and issues in addressing internalized stigma with such Veterans. Information gleaned in these qualitative interviews will form the basis of the investigators' adaption of the ESS intervention to specifically address the needs of Veterans with PTSD. In Phase II, the investigators will pilot-test ESS-P with Veterans who have PTSD, to evaluate the feasibility and acceptability of the intervention. In addition, the investigators will preliminarily estimate the effects of ESS-P through comparison to a control group receiving only an informational brochure on internalized stigma associated with PTSD. These feasibility, implementation and pilot outcome data will be used to further refine the intervention, towards the goal of conducting a future larger scale study of ESS-P within the VA system.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of PTSD
* age between 18 and 70
* participation in mental health services at the VAMHCS
* sufficient clinical stability to participate

Exclusion Criteria:

* a diagnosis of serious mental illness

  * schizophrenia/schizoaffective disorder
  * bipolar disorder
  * major depression with psychotic features
* participation in the Phase I qualitative study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Drapalski, PhD, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drapalski AL, Aakre J, Brown CH, Romero E, Lucksted A. The Ending Self-Stigma for Posttraumatic Stress Disorder (ESS-P) Program: Results of a Pilot Randomized Trial. J Trauma Stress. 2021 Feb;34(1):69-80. doi: 10.1002/jts.22593. Epub 2020 Oct 15. PMID 33058277

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ending Self-Stigma for PTSD | Enhanced Treatment as Usual
Started | 29 | 28
Completed | 24 | 18
Not Completed | 5 | 10
Not completed — Lost to Follow-up | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ending Self-Stigma for PTSD | Enhanced Treatment as Usual | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (13.0) | 55.5 (8.5) | 53.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Internalized Stigma of Mental Illness Inventory (Internalized Stigma)
Description: The Internalized Stigma of Mental Illness Inventory was used to measure of internalized or self-stigma. A total score is calculated by taking an average of the responses on the items (range=1 to 4). Higher total scores indicate greater internalized stigma.
Time Frame: Basline and Post Treatment (~3 1/2 months)
Population: Number analyzed in the rows differ from overall because 5 participants in the ESS-P and 10 in the eTAU did not complete the post-treatment assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ending Self-Stigma for PTSD | Enhanced Treatment as Usual
Number analyzed (Participants) | 29 | 28
units on a scale
  Baseline | 2.5 (0.6) | 2.6 (0.5)
  Post-treatment: number analyzed (Participants) | 24 | 18
  Post-treatment | 2.1 (0.6) | 2.5 (0.7)

2. Secondary Outcome: General Self-Efficacy
Description: The General Self-Efficacy subscale of Sherer's Self-Efficacy Scale was used to measure participant's general beliefs or expectations about their abilities. A total score is calculated by summing the responses on the items (range= 17-85). Higher score indicate greater general self-efficacy.
Time Frame: Baseline and Post Treatment (~3 1/2 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Enhanced Treatment as Usual: The comparison condition will consist of providing a pamphlet that discusses societal stigma and internalized stigma, and provides resources to help combat the effects of both. Participants will be given the informational pamphlet and study staff will discuss its content with the participant.
  .
Arm/Group | Ending Self-Stigma for PTSD | Enhanced Treatment as Usual
Number analyzed (Participants) | 29 | 28
units on a scale
  Baseline | 54.7 (11.7) | 55.4 (9.6)
  Post-Treatment: number analyzed (Participants) | 24 | 18
  Post-Treatment | 57.6 (13.3) | 53.1 (13.0)

3. Secondary Outcome: Social Self-Efficacy
Description: The Social Self-Efficacy subscale of Sherer's Self-Efficacy Scale was used to measure participant's beliefs or expectations about their abilities with regards to social interactions/relationships. A total score is calculated by summing the responses on the items (range= 5-30). Higher score indicate greater social self-efficacy.
Time Frame: Baseline and Post Treatment (~3 1/2 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ending Self-Stigma for PTSD | Enhanced Treatment as Usual
Number analyzed (Participants) | 29 | 28
units on a scale
  Baseline | 16.1 (4.9) | 15.6 (4.7)
  Post-Treatment: number analyzed (Participants) | 24 | 18
  Post-Treatment | 18.2 (4.5) | 15.7 (5.8)

ADVERSE EVENTS:
Time Frame: Adverse data were collected during their participation in the study (approximately 5 months)
Arm/Group | Ending Self-Stigma for PTSD | Enhanced Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes